CLINICAL TRIAL: NCT06071221
Title: Improving the Mental Health of Home Health Aides: A Pilot Randomized Controlled Trial
Brief Title: Improving the Mental Health of Home Health Aides
Acronym: MINDSET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-02024420
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Issue
Keywords: behavioral health intervention; home health aide; depressive symptoms; peer coaching; stress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living Healthy educational program + Peer Coaching (Experimental): Home Health Aides (HHAs) will receive educational content via the CareConnect application, an eLearning mobile platform that provides educational courses for HHA certification and keeps track of their service hours to maintain NYS compliance. HHAs in this intervention arm will receive the 8-session adapted Living Healthy program via CareConnect over 3 months. Each HHA will be paired with a trained Peer Coach participant who will work through the structured program with the HHA.
  Interventions: Behavioral: Living Healthy educational program + peer coaching
- Living Healthy educational program (Active Comparator): Home Health Aides (HHAs) in the attention control arm will receive an 8-session CareConnect delivered general health program (covering topics distinct from the Living Healthy intervention) that is strictly informational without any elements of CBT.
  Interventions: Behavioral: Living Healthy educational program

INTERVENTIONS:
Behavioral: Living Healthy educational program + peer coaching — The Living Healthy intervention is an 8-session health education program with cognitive behavioral training (CBT) techniques. For those in the interventional arm, the Living Healthy intervention program will be delivered by trained peer coaches by telephone or Zoom over 3 months. In this study, trained peer coaches are trained home health aides themselves. Informed by social cognitive theory (SCT), peer coaches train participants on cognitive behavior techniques and empower participants to adopt positive health behaviors through personalized goal setting, motivational interviewing, and peer modeling. Each content-based session incorporates principles of CBT, teaching participants to recognize and modify negative thinking and modifying outcome expectations through self-monitoring, reflection, and practice.
  Arms: Living Healthy educational program + Peer Coaching
Behavioral: Living Healthy educational program — Participants assigned to receive health education alone will be asked to read health education (online; covering aspects of the Living Healthy program) which corresponds to a weekly topic about health. They will be called by a research assistant each week to prompt them to do this and answer any questions they might have about the materials.
  Arms: Living Healthy educational program

SUMMARY:
The goal of this study is to improve the mental health of home health aides, a workforce that provides care for adults at home but whose own health has been historically poor. The main questions the study aims to answer are:

* Will a health program called Living Healthy, which provides health education and support with positive thinking, be used by home health aides and do they like it?
* Does Living Healthy actually improve home health aides' mood compared to what they usually do to take care of themselves?

Participants in the study will get an 8-week health program called Living Healthy over 3 months. Some of the participants will also have a 'peer coach' who is another home health aide who's been trained to help them with the program and learn some ways to feel better.

The study will compare the experiences of home health aides who get Living Healthy plus a peer coach with those who only get the Living Healthy program.

DETAILED DESCRIPTION:
The overall goal of the proposed project is to improve the mental health of home health aides, one of the fastest growing sectors of the healthcare industry, comprised predominantly of middle-aged women of color with high levels of stress, depressive symptoms, and emotional exhaustion. Improving home health aides' mental health and well-being is not only critical to their own longevity as a workforce, but it has the potential to improve the health of the patients for whom they care. The investigators propose adapting the Living Healthy intervention, a 8-session peer coach-delivered cognitive behavioral therapy program on healthy habits, to the home health aide workforce and pilot testing it. The specific aim of this study is to conduct a 2-arm pilot randomized control trial among 100 home health aides (intervention arm: 50; enhanced usual care arm: 50) to evaluate the feasibility, acceptability, and preliminary effectiveness of the intervention compared to enhanced usual care (education on healthy habits alone). The primary hypothesis is that the intervention will be feasible (>80% of aides will complete the program) and acceptable (>90% of aides will report high levels of satisfaction). The secondary hypothesis is that participants who receive the intervention arm will experience fewer depressive symptoms at follow-up, compared to those in the control arm. Most of the study will be conducted virtually, while initial onboarding may be in-person.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a home health aide
* Speak English or Spanish
* ≥ 18 years of age
* Have mild depressive symptoms (Personal Health Questionnaire 8-item [PHQ8] scale ≥ 5 points), or other risk factors for poor mental health as assessed by the following domains including stress (Cohen's Perceived Stress 4-item scale [PSS4] ≥5) or loneliness (≥6 on the 3-item UCLA Loneliness scale).

Exclusion Criteria:

* Speak a language other than English or Spanish
* Less than 1 year of job experience as a home health aide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fidelity to study protocol (intervention arm) | at 6 months post-intervention
  Measured by the number of total meeting attendance
Fidelity to study protocol (control arm) | at 6 months post-intervention
  Measured by the number of total meeting attendance
Fidelity to session completion (intervention arm) | at 6 months post-intervention
  Measured by number of sessions completed (participants)
Fidelity to session completion (control arm) | at 6 months post-intervention
  Measured by number of sessions completed (participants)
Fidelity to study protocol (intervention) | at 6 months post-intervention
  Measured by number intervention components delivered (peer coaches)
Accrual rate | at 3 months
  Measured by the number of participants enrolled divided by the number of months the study is open to enrollment
Refusal rate | at 3 months
  Measured by the number of participants who refuse to participate divided by the number of eligible participants
Retention rate as measured by the proportion of participants who provide 6 month combined data. | at 6 month post-intervention
  Participants who discontinue the intervention (refuse phone calls) but complete the outcome assessments will be counted in the numerator for calculating retention.
Adherence to the intervention | at 6 months post-intervention
  Measured by the proportion of participants who completed three or more sessions
Acceptability | at 6 months post-intervention
  Measured by the proportion of participants responding positively to a quantitative exit survey

SECONDARY OUTCOMES:
Change in depressive symptoms from baseline compared to 6 month assessed with the PHQ-8 | From baseline to 6-month post-intervention
  The investigators will assess the change in depressive symptoms using the PHQ-8, a validated scale that assesses depressive symptoms. This scale is composed of 8 Likert-type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 24. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. Change will be measured with repeated Anova analysis.
Change in depressive symptoms from baseline compared to 6 month assessed with the PHQ-8 | From baseline to 6-month post-intervention (attention control arm)
  The investigators will assess the change in depressive symptoms using the PHQ-8, a validated scale that assesses depressive symptoms. This scale is composed of 8 Likert-type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 24. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. Change will be measured with repeated Anova analysis.

OTHER OUTCOMES:
Change in stress from baseline compared to 6 months assessed with the Cohen's Perceived Stress (PSS-4) 4-item scale | From baseline to 6-month post-intervention
  The investigators will assess the change in stress using the PSS-4, a validated scale that assesses perceived stress experienced over the prior month. This scale is composed of 4 Likert-type items with a response scale ranging from 0 (Never) to 4 (Very Often). Total score ranges from 0 to 16. Scores greater than 5 represent moderate or greater stress.
Change in loneliness from baseline compared to 6 months assessed with the UCLA Loneliness scale 3-item scale | From baseline to 6-month post-intervention
  The investigators will assess the change in loneliness using the UCLA Loneliness scale, a validated scale that assesses feelings of loneliness. This scale is composed of 3 Likert-type items with a response scale ranging from 1 (Hardly ever or never) to 3 (Often). Scores are summed and divided by 3 to provide a mean loneliness score (1-3), with higher scores indicating greater loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline R Sterling, MD, MPH, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - 1199 SEIU Home Care Industry Education Fund, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No